CLINICAL TRIAL: NCT03466060
Title: Clinical Evaluation of 3 Contact Lens Materials With 3 Solution Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6012
Record Dates: First submitted 2018-02-26; First posted 2018-03-15 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Visual Acuity, Slit Lamp Biomicroscopy (Corneal Staining Assessment)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- etafilcon A (Active Comparator): Eligible subjects were randomized to the etafilcon A lens in both eyes throughout the entire duration of the study.
  Interventions: Device: Opti-Free : RevitaLens / Clear Care : RevitaLens; Device: Opti-Free : RevitaLens / RevitaLens : Clear Care; Device: Clear Care : RevitaLens/ Opti-Free : RevitaLens; Device: Clear Care : RevitaLens / RevitaLens : Opti-Free; Device: RevitaLens : Clear Care/ Opti-Free : RevitaLens; Device: RevitaLens : Clear Care / RevitaLens : Opti-Free; Device: RevitaLens : Opti-Free / Clear Care : RevitaLens; Device: RevitaLens : Opit-Free / RevitaLens : Clear Care
- senofilcon A (Active Comparator): Eligible subjects were randomized to the senofilcon A lens in both eyes throughout the entire duration of the study.
  Interventions: Device: Opti-Free : RevitaLens / Clear Care : RevitaLens; Device: Opti-Free : RevitaLens / RevitaLens : Clear Care; Device: Clear Care : RevitaLens/ Opti-Free : RevitaLens; Device: Clear Care : RevitaLens / RevitaLens : Opti-Free; Device: RevitaLens : Clear Care/ Opti-Free : RevitaLens; Device: RevitaLens : Clear Care / RevitaLens : Opti-Free; Device: RevitaLens : Opti-Free / Clear Care : RevitaLens; Device: RevitaLens : Opit-Free / RevitaLens : Clear Care
- senofilcon C (Active Comparator): Eligible subjects were randomized to the senofilcon C lens in both eyes throughout the entire duration of the study.
  Interventions: Device: Opti-Free : RevitaLens / Clear Care : RevitaLens; Device: Opti-Free : RevitaLens / RevitaLens : Clear Care; Device: Clear Care : RevitaLens/ Opti-Free : RevitaLens; Device: Clear Care : RevitaLens / RevitaLens : Opti-Free; Device: RevitaLens : Clear Care/ Opti-Free : RevitaLens; Device: RevitaLens : Clear Care / RevitaLens : Opti-Free; Device: RevitaLens : Opti-Free / Clear Care : RevitaLens; Device: RevitaLens : Opit-Free / RevitaLens : Clear Care

INTERVENTIONS:
Device: Opti-Free : RevitaLens / Clear Care : RevitaLens — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: Opti-Free : RevitaLens / RevitaLens : Clear Care — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: Clear Care : RevitaLens/ Opti-Free : RevitaLens — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: Clear Care : RevitaLens / RevitaLens : Opti-Free — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: RevitaLens : Clear Care/ Opti-Free : RevitaLens — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: RevitaLens : Clear Care / RevitaLens : Opti-Free — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: RevitaLens : Opti-Free / Clear Care : RevitaLens — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye
Device: RevitaLens : Opit-Free / RevitaLens : Clear Care — Subjects between the ages of 18-69 will be randomized to 1 of 3 lenses. Solutions will be administered contralaterally with 1 test solution and 1 of 2 control solutions prior to the subjects' follow-up visits.
  Other Names: Right eye : left eye / right eye : left eye

SUMMARY:
This is a multi-site, randomized, double-masked, contralateral, 2 treatment x 2 period crossover, dispensing, five-visit study to gain clinical insights of the study lenses and solutions.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. Subjects must be 18-69 years of age (inclusive).
  2. Subjects must be habitual disposable hydrogel or silicone hydrogel (1-day, 2-week, or monthly replacement schedule) soft lens wearer in both eyes. Habitual is defined as at least one (1) month of contact lens wear where the lenses are worn for a minimum of six (6) hours per day and a minimum of five (5) days per week.
  3. Subjects must have best corrected visual acuity of 20/25 (Snellen or equivalent) or better in each eye.
  4. The subject's refractive sphere (vertexed) must be between -1.00 and -6.00 D in each eye.
  5. The subject's refractive cylinder must be less than or equal to -1.00 D in each eye.
  6. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
  7. Subjects must possess a functional/usable pair of spectacles and bring them to the visit (only if applicable - to the investigators discretion).
  8. Subjects must read, understand, and sign the Statement of Informed Consent.
  9. Subjects must appear able and willing to adhere to the instructions set forth in this clinical protocol.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or breast-feeding.
  2. Diabetes
  3. Any ocular or systemic allergies or disease which may interfere with contact lens wear (at the discretion of the investigator).
  4. Any systemic disease, autoimmune disease, or use of medication which may interfere with contact lens wear (at the discretion of the investigator).
  5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (eg, HIV), by self-report.
  6. Current habitual use of Restasis, Xiidra, ocular steroids, or any medication (RX or OTC) that may interfere with contact lens wear (at the discretion of the investigator).
  7. Grade 2 or greater corneal staining or conjunctival injection on the FDA scale.
  8. Clinically significant (Grade 3 or greater on the FDA scale) corneal edema, corneal vascularization, or any other abnormalities of the cornea (excluding corneal staining) which would contraindicate contact lens wear.
  9. Clinically significant (Grade 3 or greater on the FDA scale) tarsal abnormalities which might interfere with contact lens wear.
  10. Any active ocular abnormalities/conditions that may interfere with contact lens wear (at the discretion of the investigator).
  11. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology.
  12. History of any ocular or corneal surgery (eg, RK, PRK, LASIK).
  13. Habitual contact lens wear modality as extended wear.
  14. Participation in any pharmaceutical or medical device related clinical trial within 7 days prior to study enrollment.
  15. History of binocular vision abnormality or strabismus.
  16. Habitual wearers of rigid gas permeable lens within the past 3 months.
  17. Employees of investigational clinic (investigator, coordinator, and technician etc.) or family members of employees of the investigational clinic by self-report

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Southern California College of Optometry, Anaheim, California
  - University of California, Berkeley School of Optometry, Berkeley, California
  - Vue Optical Boutique, Jacksonville, Florida
  - The Ohio State University, Columbus, Ohio
  - University of Houston College of Optometry, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 130 subjects were enrolled into this study. Of those enrolled, 113 subjects were assigned and dispensed a study lens while, 15 subjects were screen failures and 2 subjects were assigned but not administered the Test article. Of those dispensed, 106 subjects completed the study while, 7 subjects were discontinued.
Pre-assignment Details: Of those that completed the study, 78 subjects completed without a major protocol deviation impacting a primary endpoint.
Groups:
- Etafilcon A-Opti-Free/Clear Care: Subjects that were dispensed the etafilcon A lens throughout the entire study and received Opti-Free in one eye during first period and Clear in one eye during second period. During both periods Revitalens was received on the contralateral eye.
- Etafilcon A-Clear Care/Opti-Free: Subjects that were dispensed the etafilcon A lens throughout the entire study and received Clear Care in one eye during first period and Opti-Free in one eye during second period. During both periods Revitalens was received on the contralateral eye.
- Senofilcon A-Opti-free/Clear Care: Subjects that were dispensed the senofilcon A lens throughout the entire study and received Opti-Free in one eye during first period and Clear Care in one eye during second period. During both periods Revitalens was received on the contralateral eye.
- Senofilcon A-Clear Care/Opti-Free: Subjects that were dispensed the senofilcon A lens throughout the entire study and received Clear Care in one eye during first period and Opti-Free in one eye during second period. During both periods Revitalens was received on the contralateral eye.
- Senofilcon C-Opti-Free/Clear Care: Subjects that were dispensed the senofilcon C lens throughout the entire study and received Opti-Free in one eye during first period and Clear Care in one eye during second period. During both periods Revitalens was received on the contralateral eye.
- Senofilcon C-Clear Care/Opti-Free: Subjects that were dispensed the senofilcon C lens throughout the entire study and received Clear Care in one eye during first period and Opti-Free in one eye during second period. During both periods Revitalens was received on the contralateral eye.
Period: Period 1
Arm/Group | Etafilcon A-Opti-Free/Clear Care | Etafilcon A-Clear Care/Opti-Free | Senofilcon A-Opti-free/Clear Care | Senofilcon A-Clear Care/Opti-Free | Senofilcon C-Opti-Free/Clear Care | Senofilcon C-Clear Care/Opti-Free
Started | 19 | 18 | 20 | 18 | 20 | 18
Completed | 19 | 16 | 17 | 17 | 20 | 18
Not Completed | 0 | 2 | 3 | 1 | 0 | 0
Not completed — Test Lens Damage | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Grade 2 Conjunctivitis | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Etafilcon A-Opti-Free/Clear Care | Etafilcon A-Clear Care/Opti-Free | Senofilcon A-Opti-free/Clear Care | Senofilcon A-Clear Care/Opti-Free | Senofilcon C-Opti-Free/Clear Care | Senofilcon C-Clear Care/Opti-Free
Started | 19 | 16 | 17 | 17 | 20 | 18
Completed | 19 | 16 | 16 | 17 | 20 | 18
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lens Handling Difficulties | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Etafilcon A: Subjects that wore the etafilcon A lens during the entire study.
- Senofilcon A: Subjects that wore the senofilcon A lens during the entire study.
- Senofilcon C: Subjects that wore the senofilcon C lens during the entire study.
- Total: Total of all reporting groups
Arm/Group | Etafilcon A | Senofilcon A | Senofilcon C | Total
Number analyzed (Participants) | 37 | 38 | 38 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.1 (9.41) | 27.7 (7.82) | 29.1 (10.52) | 28.3 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 30 | 27 | 77
  Male | 17 | 8 | 11 | 36
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 11 | 10 | 12 | 33
  Black or African American | 1 | 5 | 2 | 8
  Native Hawaiian or Other Pacific Island | 1 | 0 | 0 | 1
  White | 22 | 20 | 24 | 66
  Other | 2 | 3 | 0 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 38 | 38 | 113

OUTCOME MEASURES:

1. Primary Outcome: Subject Comfort
Description: Subjective assessment of initial comfort was conducted using Visual Analogue Scale (VAS) of comfort. VAS of comfort consists of a vertical line which represents continuous scale from 0 (extremely uncomfortable) to 100 (extremely comfortable). VAS comfort was measured at 1-min, 5-min, 45-min, and 2-hours post-fit. The average comfort score for each solution was reported. This is a contralateral crossover, subject used the revitalens solution in one eye throughout the entire study therefore there are twice as many observations for revitalens compared to the other solutions.
Time Frame: Up to 2-Hours Post Lens Fitting
Population: All subjects who successfully completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: Eyes
Groups:
- Revita- Lens: All subject eyes that wore contact lenses pre-soaked in Revita-lens solution up to 2 hours regardless of the lens type.
- Clear Care: All subject eyes that wore contact lenses pre-soaked in Clear Care solution up to 2 hours regardless of the lens type.
- Opti-Free: All subjects eyes that wore contact lenses pre-soaked in Opit-Free solution up to 2 hours regardless of the lens type.
Arm/Group | Revita- Lens | Clear Care | Opti-Free
Number analyzed (Participants) | 78 | 78 | 78
Number analyzed (Eyes) | 78 | 78 | 78
Units on a scale
  1-Minute Follow-up | 92.4 (11.74) | 92.4 (10.52) | 92.0 (10.58)
  5-Minute Follow-up | 63.0 (10.17) | 93.4 (8.90) | 92.3 (9.81)
  45 Minute Follow-up | 93.5 (9.48) | 93.7 (8.44) | 93.5 (7.96)
  2-Hour Follow-up | 94.7 (7.06) | 94.6 (7.32) | 94.3 (7.39)
Statistical Analysis 1: Comparison: Revita- Lens vs Clear Care; 1-Minute Follow-up Analysis; Test type: Superiority; bayesian multivariate hierarachical — 95% credible intervals are used to determine whether Test and Control solutions are statistically significantly different at each time point; Posterior mean difference = -2.1, 95% CI 2-sided [-6.4 to 2.3], Standard Deviation 2.23 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 2: Comparison: Revita- Lens vs Clear Care; 5-minute Follow-up Analysis; Test type: Superiority; Bayesian Multivariate Hierarchical Model — [p-value comment as in outcome 1, analysis 1]; Posertior Mean Difference = -2.5, 95% CI 2-sided [-6.8 to 1.7], Standard Deviation 2.16 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 3: Comparison: Revita- Lens vs Clear Care; 45-Minute Follolw-up Analysis; Test type: Superiority; Bayesian multivariate hierarchical model — [p-value comment as in outcome 1, analysis 1]; Posterior Mean Difference = -2.7, 95% CI 2-sided [-6.9 to 1.5], Standard Deviation 2.10 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 4: Comparison: Revita- Lens vs Clear Care; 2-Hour Follow-up Analysis; Test type: Superiority; Bayesian Multivariate Heirarchical Model; Posterior Mean Difference = -2.5, 95% CI 2-sided [-6.5 to 1.4], Standard Deviation 2.01 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 5: Comparison: Revita- Lens vs Opti-Free; 1-Minute Follow-up Analysis; Test type: Superiority; Bayesian Multivariate Heirarchical Model; Posterior Mean Difference = -1.1, 95% CI 2-sided [-5.8 to 3.1], Standard Deviation 2.28 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 6: Comparison: Revita- Lens vs Opti-Free; 5-Minute Follow-up Analysis; Test type: Superiority — 95% credible intervals are used to determine whether Test and Control solutions are statistically significantly different at each time point; Bayesian Multivariate Heirarchical Model; Posterior Mean Difference = -0.7, 95% CI 2-sided [-5.0 to 3.6], Standard Deviation 2.20 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 7: Comparison: Revita- Lens vs Opti-Free; 45-Minute Follow-up Analysis; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 6]; Bayesian Multivariate Hierarchical Model; Posterior Mean Difference = -2.0, 95% CI 2-sided [-6.4 to 2.3], Standard Deviation 2.16 — Posterior mean difference was calculated as Test-Control
Statistical Analysis 8: Comparison: Revita- Lens vs Opti-Free; 2-Hour Follow-up Analysis; Test type: Superiority; Bayesian Mutlivariate Hiearachical Model — [p-value comment as in outcome 1, analysis 1]; Posterior Mean Difference = -1.5, 95% CI 2-sided [-5.8 to 2.5], Standard Deviation 2.10 — Posterior mean difference was calculated as Test-Control

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 5-weeks per subject.
Groups:
- Etafilcon A - Revitalens: Subjects that wore the etaiflcon A lens throughout the entire duration of the study and the revitalens solution in at least one eye throughout the entire study.
- Etafilcon A - Clear Care: Subjects that wore the etaiflcon A lens throughout the entire duration of the study and the Clear Care solution in one duringeither period 1 or period 2 during the study.
- Etafilcon A- Optifree: Subjects that wore the etaiflcon A lens throughout the entire duration of the study and the OPti-Free solution in one duringeither period 1 or period 2 during the study.
- Senofilcon A - Revitalens: Subjects that wore the senfilcon A lens throughout the entire duration of the study and the revitalens solution in at least one eye throughout the entire study.
- Senofilcon A - ClearCare: Subjects that wore the senofilcon A lens throughout the entire duration of the study and the Clear Care solution in one duringeither period 1 or period 2 during the study.
- Senofilcon A - Opti-Free: Subjects that wore the senofilcon A lens throughout the entire duration of the study and the Opti-Free solution in one duringeither period 1 or period 2 during the study.
- Senofilcon C- Revitalens: Subjects that wore the senofilcon C lens throughout the entire duration of the study and the revitalens solution in at least one eye throughout the entire study.
- Senofilcon C - ClearCare: Subjects that wore the senofilcon C lens throughout the entire duration of the study and the Clear Care solution in one duringeither period 1 or period 2 during the study.
- Senofilcon C - OptiFree: Subjects that wore the senofilcon C lens throughout the entire duration of the study and the Opti-Free solution in one duringeither period 1 or period 2 during the study.
Arm/Group | Etafilcon A - Revitalens | Etafilcon A - Clear Care | Etafilcon A- Optifree | Senofilcon A - Revitalens | Senofilcon A - ClearCare | Senofilcon A - Opti-Free | Senofilcon C- Revitalens | Senofilcon C - ClearCare | Senofilcon C - OptiFree
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38 | 0/38

LIMITATIONS AND CAVEATS:
This is a contralateral crossover, subject used the revitalens solution in one eye throughout the entire study therefore there are twice as many observations for revitalens compared to the other solutions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03466060/Prot_SAP_000.pdf